CLINICAL TRIAL: NCT01625442
Title: Effect of Crocus Sativus (Saffron) and Berberis Vulgaris (Barberry Fruit) on Metabolic Syndrome
Brief Title: Crocus Sativus (Saffron) and Berberis Vulgaris (Barberry Fruit) in Metabolic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Birjand University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3132012; 3132012n (Other: birjand university of medical sciences)
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Metabolic Syndrome; Hypercholesterolemia; Hypertriglyceridemia; Hyperglycemia
Keywords: Metabolic syndrome; hypercholesterolemia; hypertriglyceridemia; hyperglycemia
MeSH Terms: conditions — Metabolic Syndrome; Hypercholesterolemia; Hypertriglyceridemia; Hyperglycemia | interventions — crocin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Saffron (Active Comparator): Saffron treatment group received saffron tablets daily for 45 days
  Interventions: Drug: Saffron tablet
- Barberry (Active Comparator): Barberry group received barberry tablets daily for 45 days
  Interventions: Drug: Barberry tablet
- Placebo (Placebo Comparator): Placebo group received placebo tablets daily for 45 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saffron tablet — Saffron tablets 100 mg
  Other Names: crocin
  Arms: Saffron
Drug: Barberry tablet — Barberry tablets 200 mg
  Arms: Barberry
Drug: Placebo — Placebo tablets received daily for 45 days
  Arms: Placebo

SUMMARY:
The metabolic syndrome is associated with increased risk of cardiovascular disease and diabetes mellitus. The age-adjusted prevalence of the metabolic syndrome in the United States is 34% for men and 35% for women. Emerging alternative medicine worldwide led investigators to evaluate the efficacy of Crocus sativus (Saffron) and Berberis Vulgaris (barberry fruit) in treatment of metabolic syndrome. Serum total cholesterol, serum LDL cholesterol, serum HDL cholesterol, serum triglyceride, Fasting Blood Sugar and hematocrit measured before and after 45 days of treatment.

DETAILED DESCRIPTION:
In a randomized, placebo controlled, single-blind , efficacy trial with three treatment arms the investigators randomly assigned 105 patients with metabolic syndrome to receive barberry juice, saffron juice or placebo tablet.

The aim was to evaluate the efficacy of Crocus sativus (Saffron) and Berberis Vulgaris (barberry fruit) in treatment of metabolic syndrome. The metabolic syndrome (syndrome X, insulin resistance syndrome) consists of a constellation of metabolic abnormalities that confer increased risk of cardiovascular disease (CVD) and diabetes mellitus (DM). The major features of the metabolic syndrome include central obesity hypertriglyceridemia, low HDL cholesterol, hyperglycemia, and hypertension. Based on data from the National Health and Nutrition Examination Survey (NHANES) III, the age-adjusted prevalence of the metabolic syndrome in the United States is 34% for men and 35% for Women. Review of literature revealed anti-inflammatory, radical-scavenging, antioxidant, cytoprotective, beneficial cardiovascular and neural system effects for saffron, potential use for treatment of hypertension, tachycardia and some neuronal disorders, such as epilepsy and convulsion, antihypertensive and vasodilatory activities. Barberry has promising and selective anti-cancer activities, beneficial effects in atherosclerosis, arthritis, coronary heart disease and hepatitis, hypotensive property and to promote immunity, prevention of insulin resistance and related diseases, neuroprotective, hypolipidemic and antioxidant properties for saffron in animal models.

ELIGIBILITY:
Inclusion Criteria:

* waist circumference of ≥ 94 cm (males) or ≥ 80 cm (females) plus any two of the following:
* blood pressure ≥ 130/85 or taking antihypertensive medication,
* fasting plasma glucose (FPG) > 100 mg/dL,
* serum triglycerides (TG) > 150 mg/dL,
* high-density lipoprotein (HDL) < 40 mg/dL in men,and < 50 mg/dL in women-

Exclusion Criteria:

* using insulin or glucose sensitizing medication
* preexisting cardiovascular disease
* psychiatric problems
* non-compliance of patients
* not presenting at times determined for treatment and evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 732 (Actual)
Dates: Start 2010-01; Primary Completion 2011-07 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Serum LDL cholesterol | after 45 days of treatment
  Serum LDL cholesterol after 45 days of treatment in three study groups

SECONDARY OUTCOMES:
Serum total cholesterol | after 45 days of treatment
  Serum total cholesterol after 45 days of treatment in three study groups
serum HDL cholesterol | after 45 days of treatment
  serum HDL cholesterol after 45 days of treatment in three study groups
serum triglyceride | after 45 days of treatment
  serum triglyceride after 45 days of treatment in three study groups
Fasting Blood Sugar | after 45 days of treatment
  Fasting Blood Sugar after 45 days of treatment in three study groups
Hematocrit | after 45 days of treatment
  Hematocrit measured after 45 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tayyebeh Kermani, Ph.D., Principal Investigator — Assistant proffessor of anatomy; Maryam Navabzadeh, M.D., Study Director — Traditional iranian medicine specialist; Gholamreza Sharifzadeh, M.S., Principal Investigator — Biostatistician; Javad Hadinia, B.S., Principal Investigator — Traditional iranian medicine practitioner; Narges Saffari, B.S., Principal Investigator — Health technician; Mohammad Khodashenas Roudsari, M.D., Study Chair — Assistant proffessor of internal medicine
Locations (1):
- Birjand University of medical sciences, Birjand, South Khorasan Province, Iran